CLINICAL TRIAL: NCT04354246
Title: A Phase 1 Study of The Safety and Tolerability of COM902 in Subjects With Advanced Malignancies
Brief Title: COM902 (A TIGIT Inhibitor) in Subjects With Advanced Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Compugen Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CPG-02-101
Record Dates: First submitted 2020-04-15; First posted 2020-04-21 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Advanced Cancer; Ovarian Cancer; Lung Cancer; Colon Cancer; Plasma Cell Neoplasm; Multiple Myeloma; HNSCC; Microsatellite Stable Colorectal Carcinoma; MSS-CRC
Keywords: TIGIT antibody; PVRIG antibody; COM701; Low Fc-effector function; Pembrolizumab
MeSH Terms: conditions — Ovarian Neoplasms; Lung Neoplasms; Colonic Neoplasms; Neoplasms, Plasma Cell; Multiple Myeloma; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- COM902 monotherapy dose escalation. (Experimental): Monotherapy dose escalation. COM902 monotherapy administered IV every 3 weeks in sequential dose escalation. Up to 7 dose escalation cohorts may be evaluated until a maximum tolerated dose or recommended dose for expansion (RDFE) is identified.
  Interventions: Drug: Dose escalation: COM902 monotherapy.
- Dual combination (COM902 + COM701) for evaluation of safety/tolerability (both at RDFE). (Experimental): COM902 will be combined with COM701 for evaluation of safety and tolerability. All study drugs will be administered IV every 3 weeks.
  Interventions: Combination Product: Evaluation of safety/tolerability: COM902 in combination with COM701 (both at the RDFE)
- COM902 monotherapy cohort expansion at RDFE. (Experimental): COM902 monotherapy at the RDFE - in subjects with multiple myeloma. COM902 will be administered IV every 3 weeks.
  Interventions: Drug: Cohort expansion: COM902 (RDFE) monotherapy.
- COM902 + COM701 combination cohort expansion both at RDFE. (Experimental): COM902 + COM701 (both at the RDFE) evaluated in subjects with select tumor types who have exhausted standard of care treatment: HNSCC, CRC (MSS), NSCLC. All study drugs will be administered IV every 3 weeks.
  Interventions: Drug: Cohort expansion: COM902 in combination with COM701 (both at the RDFE).
- MSS-CRC Triplet combination (COM902 + COM701 + Pembrolizumab). (Experimental): Triplet combination of COM902 + COM701 + Pembrolizumab evaluated in subjects with MSS-CRC. All study drugs will be administered IV every 3 weeks.
  Interventions: Combination Product: Cohort expansion: Triplet combination of COM902 + COM701 + Pembrolizumab.
- Platinum resistant ovarian cancer Triplet combination (COM902 + COM701 + Pembrolizumab). (Experimental): Triplet combination of COM902 + COM701 + Pembrolizumab evaluated in subjects with PROC. All study drugs will be administered IV every 3 weeks.
  Interventions: Combination Product: Cohort expansion: Triplet combination of COM902 + COM701 + Pembrolizumab.

INTERVENTIONS:
Drug: Dose escalation: COM902 monotherapy. — COM902 monotherapy administered IV every 3 weeks in sequential dose escalation doses in cohorts of subjects.
  Arms: COM902 monotherapy dose escalation.
Combination Product: Evaluation of safety/tolerability: COM902 in combination with COM701 (both at the RDFE) — Both study drugs will be evaluated at the RDFE for assessment of safety and tolerability. All study drugs will be administered IV every 3 weeks.
  Arms: Dual combination (COM902 + COM701) for evaluation of safety/tolerability (both at RDFE).
Drug: Cohort expansion: COM902 (RDFE) monotherapy. — COM902 monotherapy (RDFE) in subjects with multiple myeloma. COM902 will be administered IV every 3 weeks.
  Arms: COM902 monotherapy cohort expansion at RDFE.
Drug: Cohort expansion: COM902 in combination with COM701 (both at the RDFE). — COM902 in combination with COM701 (both at RDFE) in subjects with select tumor types who have exhausted standard treatment - HNSCC, CRC (MSS), NSCLC. All study drugs will be administered IV every 3 weeks.
  Arms: COM902 + COM701 combination cohort expansion both at RDFE.
Combination Product: Cohort expansion: Triplet combination of COM902 + COM701 + Pembrolizumab. — Triplet combination of COM902 + COM701 + Pembrolizumab administered IV every 3 weeks.
  Arms: MSS-CRC Triplet combination (COM902 + COM701 + Pembrolizumab).; Platinum resistant ovarian cancer Triplet combination (COM902 + COM701 + Pembrolizumab).

SUMMARY:
Phase 1 open label sequential dose escalation and cohort expansion study evaluating the safety, tolerability and preliminary antitumor activity of COM902 as monotherapy and in combination with COM701 in subjects with advanced malignancies.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects with histologically/cytologically confirmed advanced malignancy (solid tumor) who must have exhausted all available standard therapy, or not a candidate for standard therapy.
* Subject is able to provide written, informed consent before initiation of any study related procedures, and is able, in the opinion of the investigator, to comply with all the requirements of the study.
* Subject has Eastern Cooperative Oncology Group (ECOG) performance status 0-1.

For Triplet combination MSS-CRC:

* Histologically confirmed adenocarcinoma of the colon/rectum
* Stage IV disease
* MSS-CRC status by an FDA approved test
* Disease progression with no more than 3 prior lines of treatment including fluroropyrimidines, irinotecan, and oxaliplatin

For Triplet combination ovarian cancer:

* Advanced epithelial ovarian, fallopian tube, or primary peritoneal carcinoma
* Platinum resistant ovarian cancer (PROC) defined as disease recurrence < 6 months after completion of a platinum-containing regimen: Patients with primary platinum refractory disease are ineligible. Primary platinum refractory disease is defined as progression of disease prior to completion of 1st line platinum therapy or immediately following (≤ 3 months following last date of chemotherapy)
* Received ≤3 prior lines for PROC; maintenance bevacizumab or PARP are not included as a line of therapy
* Subjects who have received PARP inhibitor therapy are eligible

Key Exclusion Criteria:

* Prior treatment with a TIGIT inhibitor.
* Prior treatment with an inhibitor of PVRIG
* Symptomatic interstitial lung disease or inflammatory pneumonitis.
* History of immune-related events that required immunotherapy treatment discontinuation

For Triplet combination expansion cohorts (MSS-CRC and PROC): Prior treatment with an anti-PD-1/PD-L1/2, anti-CD96 antibody, anti-OX-40 antibody, anti-CD137 antibody, anti-LAG3, anti-TIM3, anti-CTLA4 antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-03-31 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The safety and tolerability of COM902 monotherapy and in combination with COM701. | DLT evaluation window in the 1st cycle (21 Days).
  Incidence of subjects with Adverse Events (AEs) as per CTCAE v5.0 and Dose-Limiting Toxicities (DLTs).
To identify the maximum tolerated dose (MTD) and/or recommended dose for expansion of COM902 monotherapy and in combination with COM701. | 18 months.
  Evaluation of a dose of COM902 monotherapy and in combination with COM701 that is well tolerated by subjects.
To characterize the pharmacokinetic (PK) profile of COM902 as monotherapy and in combination with COM701. | 18 months.
  Evaluation of parameters of COM902 monotherapy or in combination with COM701 exposure such as Maximum Plasma Concentration [Cmax]).
Evaluation of safety and tolerability of the Triplet combination (COM902 + COM701 + Pembrolizumab). | 18 months.
  Incidence of subjects on the Triplet combination (COM902 + COM701 + Pembrolizumab) with Adverse Events (AEs) per CTCAE v5.0.
Evaluation of the PK profile of the Triplet combination (COM902 + COM701 + Pembrolizumab). | 18 months.
  Evaluation of PK parameters e.g., Cmax.
Evaluation of the PK profile of the Triplet combination (COM902 + COM701 + Pembrolizumab). | 18 months.
  Evaluation of PK parameters e.g., AUC.

SECONDARY OUTCOMES:
To characterize immunogenicity of COM902 monotherapy and in combination with COM701. | 18 months.
  Evaluation of anti drug antibody to COM902 (monotherapy) or COM902, COM701 when administered in combination.
To characterize the immunogenicity of the Triplet combination (COM902 + COM701 + Pembrolizumab). | 18 months.
  Evaluation of antidrug antibody to COM902, COM701.

OTHER OUTCOMES:
Evaluation of the preliminary antitumor activity of COM902 as monotherapy and in combination with COM701. | 24 months.
  An assessment of preliminary antitumor activity eg ORR with COM902 monotherapy and COM902 in combination with COM701.
Preliminary antitumor activity of the triplet combination (COM902 + COM701 + Pembrolizumab). | 24 months
  Assessment of preliminary antitumor activity e.g., ORR.

CONTACTS AND LOCATIONS:
Overall Officials: COM902 Study Director COM902 Study Director, Study Director — Compugen Ltd
Locations (9):
- United States (9):
  - Florida Cancer Specialists, Sarasota, Florida
  - Massachusetts General Hospital., Boston, Massachusetts
  - START Midwest., Grand Rapids, Michigan
  - The Ohio State University Comprehensive Cancer Center., Columbus, Ohio
  - The University of Tennessee WEST Cancer Center., Memphis, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson Cancer Center., Houston, Texas
  - The START Center for Cancer Care., San Antonio, Texas
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No